CLINICAL TRIAL: NCT06311630
Title: Comparative Study of Analgesic Effect of Ultrasound Guided PENG Block With FEMORAL NERVE BLOCK in Patients With Hip Fracture Presenting to Emergency Department
Brief Title: Comparative Study of Analgesic Effect of Ultrasound Guided PENG Block vs FEMORAL BLOCK in Hip Fracture
Status: Recruiting | Type: Observational
Sponsor: Jubilee Mission Medical College and Research Institute (Other)
Responsible Party: Principal Investigator, Dr. Jogi Varghese, Junior resident, Jubilee Mission Medical College and Research Institute
Other Study IDs: 65/23/IEC/JMMC&RI
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Hip Fracture
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To study the analgesic effect of ultrasound guided PENG Block vs Femoral nerve block in patients with Hip fracture presenting to Emergency department

DETAILED DESCRIPTION:
comparative study of analgesic effect of ultrasound guided PENG block vs femoral nerve block in patients presenting to emergency department

ELIGIBILITY:
Inclusion Criteria:

* Adults more than or equal to 18 yrs with Hip fracture
* patients who consent for procedure

Exclusion Criteria:

* history of allergy to local anaesthetics
* pregnant or lactating women
* infection or burns at injection site
* patients with polytrauma
* patients with hemodynamic instability
* patients with low GCS
* patients on anticoagulant or hematological disorders
* injuries with neurovascular compromise on affected limb
* patients with distorted anatomy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients with Hip fracture presenting to Emergency department
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-05-20 (Actual); Primary Completion 2025-01-20 (Estimated); Study Completion 2025-03-20 (Estimated)

PRIMARY OUTCOMES:
Comparative Study of Analgesic Effect of Ultrasound Guided PENG Block With FEMORAL NERVE BLOCK in Patients With Hip Fracture as assessed by NRS pain scoring scale by patient | 1 hour
  To study the analgesic effect of peng block vs Femoral nerve block in patients with Hip fracture by NRS (NUMERIC RATING SCALE FROM 0-10) WITH 0 MEANING NO PAIN AND 10 MEANING SEVERE PAIN

SECONDARY OUTCOMES:
Time taken for each technique | 1 hour
  Time taken for thr each procedure
Time taken for adequate analgesia | 1hour
  To study time taken for analgesic effect after procedure
Incidence of complications | 7 days
  To look for any immediate and late complications
To note if rescue analgesic is required | 1 hour
  To note if opioids are required as rescue analgesia

CONTACTS AND LOCATIONS:
Overall Officials: Jogi Varghese, MBBS, Principal Investigator
Locations (1):
- Jubilee mission medical College and research centre, Thrissur, Kerala, India

IPD SHARING:
Plan to Share IPD: No